CLINICAL TRIAL: NCT06240195
Title: Biomarkers of Efficacy and Tolerability of Sacituzumab-Govitecan in the Treatment of Patients With Triple-negative Breast Cancer in the Metastatic Phase: Prospective Multicenter Real-world Study
Acronym: BIO-PROSA
Status: Recruiting | Type: Observational
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Ospedale Sandro Pertini, Roma (Other); Catholic University of the Sacred Heart (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Campus Bio-Medico University (Other); Azienda Policlinico Umberto I (Other); San Giovanni Addolorata Hospital (Other); Ospedale "SS Annunziata", Chieti (Unknown); Ospedale "Gaetano Bernabeo" , Ortona (Unknown); Hospital San Pietro Fatebenefratelli (Other); presidio Ospedaliero santo spirito in Sassia, Roma (Unknown); Ospedale di Belcolle - Viterbo (Unknown)
Responsible Party: Sponsor
Other Study IDs: RS1814/22
Record Dates: First submitted 2024-01-12; First posted 2024-02-02 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue (where possible both primary and metastatic) and on circulating plasma collected at two separate time points (T0 and T1).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with metastatic triple-negative breast cancer treated with sacituzumab govitecan: The availability of at least one tumor tissue sample to be transferred to the coordinating center will be essential for enrollment in the study. For patients for whom a new sampling is scheduled biopsy of the tumor (primary or metastasis) as per clinical practice, the feasibility of the development will be assessed tumor organoids and the execution of single-cell sequencing on tumor tissue. In these cases, the order of priority in dividing the sampled tissue will be: sufficient quota to carry out the histological examination that will have to be carried out naturally confirm the diagnosis of triple-negative breast cancer. Quota to be prepared as a fresh preparation for the two experiments of feasibility indicated above; quota to be considered as a second sample, to be analyzed at the end of the study.
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Collection of data relating to the effectiveness of sacituzumab govitecan and evaluation in a real-world context and planned research of predictive biomarkers of efficacy/tolerability

SUMMARY:
Observational, prospective, multicenter study. Collection of data relating to the effectiveness of sacituzumab govitecan SG, in a real-world context and planned research of predictive biomarkers of efficacy/tolerability carried out on multiple platforms at the center coordinator.

DETAILED DESCRIPTION:
Identification and inclusion in the study of patients affected by metastatic triple-negative breast cancer mTNBC, treated with sacituzumab govitecan SG as indicated at the participating centers.

Histological and biomolecular characteristics will be evaluated both on the tumor at diagnosis and on tissue resulting from biopsy of the metastatic site, where available. Otherwise, the analyzes will come anyway carried out on the most recent and available tumor tissue, whether deriving from primary tumor or site metastatic.

The search for biomarkers predictive of efficacy/tolerability will be carried out on tumor tissue (where possible both primary and metastatic) and on circulating plasma collected at two separate time points (T0 and T1).

Biomolecular characterization on the biological material of the enrolled patients (tumor tissue and plasma) will be carried out at the end of the study.

The feasibility of organoid development and single-cell sequencing will be evaluated on a small subgroup of patients, among those enrolled at the coordinating center, considering the need for tumor tissue prepared fresh for both methods.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Histological diagnosis of TNBC;
* Locally advanced unresectable or metastatic disease;
* Indication for treatment with SG in monotherapy according to clinical practice (patients pre-treated with at least two lines of systemic therapy, of which at least one in an advanced stage);
* Availability of at least one tumor tissue sample (from primary tumor or metastasis) to be sent to the coordinating center (IRE);
* Written informed consent;
* Availability to comply with the procedures established by the protocol, according to the methods and times described.

Exclusion Criteria:

* Patients with a history of other malignancies;
* Contraindications to the use of sacituzumab govitecan SG;
* Untreated and/or clinically unstable (symptomatic) brain metastases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic triple-negative breast cancer treated with socituzumab govitecan as indicated, with at least one sample of tumor tissue available.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-01-17 (Estimated); Study Completion 2025-06-17 (Estimated)

PRIMARY OUTCOMES:
Biomolecular investigations conducted on multiple platforms | 30 months
  Identify the predictive factors of the efficacy of sacituzumab govitecan in terms of PFS through biomolecular investigations conducted on multiple platforms, using tumor tissue (where possible both primary and metastatic) and peripheral blood, circulating plasma collected at two separate time points (T0 and T1) of mTNBC patients treated in the real-world setting.

SECONDARY OUTCOMES:
PFS in patients. | 30 months
  Assess any differences in terms of PFS in patients treated in second line compared to patient treated in lines subsequent to the second. Evaluate the dynamics of quantitative variation over time of any circulating microRNAs predictive of efficacy and tolerability. Evaluate the differences in any predictive biomarkers of efficacy/tolerability, tissue and/or circulating, in patients treated in second line vs patients treated in subsequent lines. Assess any differences in PFS in relation to: previous treatment(s) in the early setting and metastatic, disease sites, dose reductions/treatment discontinuation.
Tolerability of the treatment | 30 months
  Evaluate the tolerability of the treatment in terms of adverse events, defined according to Common Terminology Criteria for Adverse Events (CTCAE, v. 5) and identify factors predictive of toxicity. Evaluate objective response rate (ORR) and overall survival (OS). Assess the variation in any biomarkers of efficacy in primary tumor tissue vs. tissue from metastatic localization (in cases where both samples are available). Select a small subgroup of patients from whose tumor tissue to develop organoids will be treated with SG, and on which potential will be quantified longitudinally over time biomarkers of response to treatment.
Development of organoids | 30 months
  Select a small subgroup of patients from the tumor tissue for single cell testing RNA sequencing to compare with data from bulk RNA sequencing to study the microenvironment tumoral.

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Vici, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
The Sponsor is the exclusive owner of all data and information arising from the study, including results, discoveries, know-how and the like.